CLINICAL TRIAL: NCT01761929
Title: A Phase II Study on the Toxicity and Efficacy of a Normal Tissue Tolerance Adapted, 5 Fraction Stereotactic Body Radiation Therapy (SBRT) Regimen, for Extra-Cranial Oligometastases
Brief Title: 5 Fraction Stereotactic Body Radiation Therapy for Oligometastases Regimen, for Extra-Cranial Oligometastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB '11-0886-C'
Record Dates: First submitted 2012-02-27; First posted 2013-01-07 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Solid Tumors With Oligometastatic Spread
Keywords: oligometastatic; oligometastases; stereotactic body radiotherapy; radiation therapy; Oligometastasis; Stereotactic ablative body; radiotherapy
MeSH Terms: interventions — MAX protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Body Radiation Therapy (Experimental): All patients will be treated with SBRT 1-2 weeks after radiotherapy planning scans. Therapy will be given once daily, over 5 consecutive working days according to standard practice.
  Interventions: Radiation: Radiation: 50Gy in 5 fr (max) to 25 Gy in 5 fr (min). Dose adapted to deliver the highest dose level while respecting normal tissue tolerance

INTERVENTIONS:
Radiation: Radiation: 50Gy in 5 fr (max) to 25 Gy in 5 fr (min). Dose adapted to deliver the highest dose level while respecting normal tissue tolerance — All patients will be treated with SBRT 1-2 weeks after radiotherapy planning scans. Therapy will be given once daily, over 5 consecutive working days according to standard practice.

SUMMARY:
This is a prospective Phase II study.The purpose of this study is to monitor the side effects and treatment outcomes of delivering higher doses of radiation therapy to the tumour, while limiting the dose of radiation to the normal tissues. This will be done using a 5 day treatment schedule.

The characteristics of patients whose disease remains confined to limited areas in the long term, compared with those who do not will also be described.

DETAILED DESCRIPTION:
Endpoints are to describe: the proportion of patients with local control for the index site at 1 year; the number of index lesion(s) with local control at 1 year; acute and late AEs related to SBRT; time to local progression for the index site; time to distant disease progression; symptom and QoL profile; median survival.

ELIGIBILITY:
Inclusion Criteria:

* Any solid tumors are eligible. Lymphoma, myeloma and germ cell tumors are excluded.
* Histological confirmation of neoplastic disease either from original primary or metastatic sites is required.
* Radiological diagnosis of oligometastastic metastatic disease is accepted if considered clinically acceptable. Histological confirmation is not mandatory.
* Oligometastatic disease, maximum of 5 lesions.
* At least one lesion is suitable for stereotactic body radiotherapy
* All known sites of disease have plans for local ablative management (see section management plan for definitions) within 3 months
* ECOG ≤ 2
* At least 18 yrs old

Exclusion Criteria:

* Previous radiotherapy to the intended treatment site
* Patient cannot tolerate physical set up required for SBRT
* Active bowel obstruction, if treating abdominal/pelvic site
* Chemotherapy within 2 weeks of intended radiation therapy
* Treatment plan respecting normal tissue tolerances using dose fractionation specified within the protocol cannot be achieved
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2013-03-07 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with lack of progressive disease for the index site at 1 year | 10 years
  CT will be used for evaluation of the status of the local disease at the index site.

SECONDARY OUTCOMES:
Number of index lesion(s) with lack of progressive disease at 1 year. | 10 years
  The Modified Response Evaluation Criteria for solid Tumors (RECIST) will be used. By measuring the longest diameter (LD) of the lesions, response of individual lesions and overall response will be documented.
Acute toxicity within 90 days of first fraction of radiotherapy | 10 years
  Acute toxicity will be graded according to the Common Toxicity Criteria, v4.0
Time to local progression for the index site(s) | 10 years
Time to distant disease progression (beyond known sites of oligometastases at time of study entry) | 10 years
Late toxicity occuring beyond 90 days related to SBRT. | 10 year
  Late toxicity will be graded according to the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer score.
Describe symptom profile | 10 Years
Examine radiotherapy parameters (outlined in Appendix J) for local control of index site(s) and toxicities | 10 years

OTHER OUTCOMES:
Explore pre-treatment prognostic factors derived from clinical data and correlative studies for disease free interval | 10 years
Explore pre-treatment prognostic factors derived from clinical data and correlative studies for local control of index site(s) at 1 year | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca K.S. Wong, MB ChB, Principal Investigator — University Health Network - Princess Margaret Cancer Center
Locations (1):
- University Health Network, Princess Margaret Cancer Center, Toronto, Ontario, Canada